CLINICAL TRIAL: NCT04905082
Title: Helping Oncology Patients Explore-Genomics (HOPE-Genomics) Web Tool Randomized Clinical Trial
Brief Title: HOPE-Genomics Intervention for the Improvement of Cancer Patient Knowledge of Genomics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20430; NCI-2021-03114 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20430 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma; Lung Carcinoma; Malignant Solid Neoplasm; Ovarian Carcinoma; Pancreatic Carcinoma; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Genetic Profile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (usual care) (Active Comparator): Patients receive education pamphlet about WES and have their genomics test results returned by their clinician in a typical manner.
  Interventions: Other: Best Practice; Other: Survey Administration
- Arm II (genomics test results, HOPE-Genomics) (Experimental): Patients receive their genomics test results both from their clinician and from the HOPE-Genomics tool. Patients then view HOPE-Genomics tool over 15-20 minutes after their results are available.
  Interventions: Other: Educational Intervention; Procedure: Genomic Profile; Other: Survey Administration
- Arm III (HOPE-Genomics, genomics test results) (Experimental): Patients view HOPE-Genomics tool (containing educational content) over 15-20 minutes before their sequencing results are available. Patients also receive their genomics test results both from their clinician and from the HOPE-Genomics tool.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm I (usual care)
Other: Educational Intervention — View HOPE-Genomics tool after genomic test results are available
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (genomics test results, HOPE-Genomics)
Other: Educational Intervention — View HOPE-Genomics before sequencing results are available
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm III (HOPE-Genomics, genomics test results)
Procedure: Genomic Profile — Receive genomics test results
  Other Names: genetic profile; Genome Profile; Genomic Profiling; Genomic Test; Genomic Testing
  Arms: Arm II (genomics test results, HOPE-Genomics)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effectiveness of a web-based cancer education tool called Helping Oncology Patients Explore Genomics (HOPE-Genomics) in improving patient knowledge of personal genomic testing results and cancer and genomics in general. HOPE-Genomics is a web-based education tool that teaches cancer/leukemia patients, and patients who may be at high-risk for developing cancer, about genomic testing and provide patients with information about their own genomic test results. The HOPE-Genomics tool may improve patient's genomic knowledge and quality of patient-centered care. In addition, it may also improve education and care quality for future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the efficacy of the HOPE-Genomics intervention in improving patient knowledge of genomics.

II. Test the efficacy of the HOPE-Genomics intervention in improving patient receipt of guideline-concordant care.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (USUAL CARE): Patients receive education pamphlet about whole-genome sequencing (WES) and have their genomics test results returned by their clinician in a typical manner.

ARM II (RETURN OF RESULTS ONLY): Patients receive their genomics test results both from their clinician and from the HOPE-Genomics tool. Patients then view HOPE-Genomics tool over 15-20 minutes after their results are available.

ARM III (RETURN OF RESULTS PLUS PRE-TEST EDUCATION): Patients view HOPE-Genomics tool (containing educational content) over 15-20 minutes before their sequencing results are available. Patients also receive their genomics test results both from their clinician and from the HOPE-Genomics tool.

After completion of study intervention, patients are followed up at 2 weeks, 3 and 9 months after receiving genomic test results.

ELIGIBILITY:
Inclusion Criteria:

* Are enrolled in City of Hope (COH) Institutional Review Board (IRB) 07047
* Have a diagnosis of lung, breast, colorectal, pancreatic, ovarian or prostate cancer
* Having somatic, germline or paired somatic/germline sequencing
* Are fluent in English
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Are >= 18 years old

Exclusion Criteria:

* Are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy W Gray, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) | Arm III (HOPE-Genomics, Genomics Test Results)
Started | 155 | 155 | 155
Pre-test Survey (Approximately 2-3 Days After Baseline) | 140 | 143 | 142
Ten-day Visit | 132 | 134 | 129
Three-month Survey | 121 | 122 | 122
Completed | 104 | 109 | 105
Not Completed | 51 | 46 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) | Arm III (HOPE-Genomics, Genomics Test Results) | Total
Number analyzed (Participants) | 155 | 155 | 155 | 465
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 110 | 116 | 338
  Male | 43 | 45 | 39 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 5
  Asian | 21 | 16 | 19 | 56
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 6 | 17
  White | 114 | 126 | 117 | 357
  More than one race | 11 | 5 | 6 | 22
  Unknown or Not Reported | 2 | 2 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 37 | 36 | 115
  Not Hispanic or Latino | 110 | 116 | 118 | 344
  Unknown or Not Reported | 3 | 2 | 1 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: Year] | 59 [49 to 69] | 61 [52 to 68] | 64 [52 to 72] | 61 [51 to 69]
Education [Count of Participants; unit: Participants]
  Grades 1 through 8 | 0 | 1 | 0 | 1
  Grades 9 through 11 | 4 | 0 | 2 | 6
  Grade 12 or GED | 11 | 10 | 19 | 40
  College 1 Year to 3 Years (Some College or Technical School) | 43 | 45 | 43 | 131
  College 4 years or More (College Graduate) | 45 | 48 | 44 | 137
  Master's Degree | 25 | 29 | 25 | 79
  Doctoral Degree | 13 | 14 | 18 | 45
  Unknown or Not Reported | 14 | 8 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Recall Rates of Personal Genomic Results
Description: Recall rate refers to the proportion of patients who accurately remembered whether they had undergone genetic testing, as reported in the 10-day follow-up survey. If a patient's response at the 10-day mark was unavailable, their answer from the 3-month survey was used as a substitute. This metric helps assess how well patients retained and understood information about their genetic testing experience shortly after receiving their results.
Time Frame: Up to 3 months
Population: For the primary analysis, only patients who responded to the question regarding completion of germline testing in either the 10-day or 3-month survey were included. Therefore, the number of patients analyzed differs from the total number of randomized participants.
Measure: Count of Participants; unit: Participants
Groups:
- Arm II (Genomics Test Results, HOPE-Genomics) Plus Arm III (HOPE-Genomics, Genomics Test Results): This group pools together Arm II and Arm III patients who have access to genomics test results from the HOPE-Genomics tool.
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) Plus Arm III (HOPE-Genomics, Genomics Test Results) | Arm III (HOPE-Genomics, Genomics Test Results)
Number analyzed (Participants) | 132 | 137 | 131
Participants
  Recalled Germline Testing | 89 | 82 | 83
  Not Recalled Germline Testing | 43 | 55 | 48

2. Secondary Outcome: Operationalization of Contextual Guideline Concordant Care
Description: In the primary analysis, we will assess the uptake of contextualized guideline-concordant care taking into account clinically relevant, patient specific circumstances. Will use clinical characteristics from the electronic health record (EHR) to assign each patient to clinical category for which there are discrete National Comprehensive Cancer Network (NCCN) recommendations. Using patient self-reported baseline/T1 and EHR data, following sequencing disclosure, we will create a summary genetically-guided care variable ranging from 0-100%. In the secondary analyses, will define guideline concordant as meeting >= 75% of recommended guidelines.
Time Frame: Up to 12-month period after results disclosure
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Test-related Distress
Description: The psychosocial impact of genetic testing and patient uncertainty were assessed at 10 days, 3 months and 9 months using both the adapted PAGIS Certainty Scale and the FACToR. The FACToR was a 12-item measure that included four subscales: privacy concerns, uncertainty, test-related distress, and positive experiences. The overall FACToR score is computed by summing all items after reverse scoring the positivity subscale, resulting in a total range of 0 to 48. Higher total scores indicate greater psychosocial impact, which is considered a worse outcome. The PAGIS Certainty Subscale consists of 6 items scored on a 1-6 scale, with a total range of 6-36. Higher scores reflect greater certainty and better psychological adaptation to genetic information, which is considered a positive outcome.
Time Frame: 10 days, 3 months, 9 months
Population: Only participants who answered distress-related questions were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) | Arm III (HOPE-Genomics, Genomics Test Results)
Number analyzed (Participants) | 121 | 126 | 120
scores on a scale
  FACToR Score at 10-Day: number analyzed (Participants) | 96 | 99 | 87
  FACToR Score at 10-Day | 11.07 (6.29) | 12.37 (6.82) | 11.17 (7.93)
  FACToR Score at 3-Month: number analyzed (Participants) | 79 | 87 | 75
  FACToR Score at 3-Month | 12.32 (6.83) | 13.20 (7.41) | 12.48 (7.47)
  FACToR Score at 9-Month: number analyzed (Participants) | 96 | 98 | 95
  FACToR Score at 9-Month | 12.61 (7.11) | 11.97 (6.31) | 12.19 (7.01)
  PAGIS Score at 10 Days: number analyzed (Participants) | 90 | 99 | 85
  PAGIS Score at 10 Days | 24.76 (6.74) | 24.25 (7.11) | 26.53 (6.95)
  PAGIS Score at 3 Months: number analyzed (Participants) | 83 | 89 | 75
  PAGIS Score at 3 Months | 25.11 (7.38) | 24.54 (7.23) | 26.11 (7.30)
  PAGIS Score at 9 Months: number analyzed (Participants) | 92 | 99 | 102
  PAGIS Score at 9 Months | 22.29 (7.12) | 23.11 (7.42) | 24.39 (8.34)

4. Other Pre Specified Outcome: Genetically-guided Care
Description: In exploratory analyses related to Aim 2 (i.e. receipt of contextual guideline-concordant care), will also operationalize the secondary outcome in an additional way: Categories of genetically-guided care: Will evaluate patients' receipt of 1) treatment recommended by provider based on sequencing (any/none), 2) patients' sharing of sequencing results with family members (any/none), and 3) patients' consultation with genetic counseling/ recommended specialist (any/none).
Time Frame: Up to 9 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: HOPE-Genomics Tool Usage
Description: Will analyze the web-log of user visits (e.g., number of viewing sessions, page views and use of interactive elements).
Time Frame: Up to 9 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Genomic Knowledge Score
Description: Genomic knowledge was assessed using a modified 35-item instrument comprising three subscales: cancer genomics knowledge, understanding of the use of genetic testing results in cancer care, and germline sequencing knowledge. Overall knowledge scores were calculated for patients who completed more than half of the items in the full measure. Each score was expressed as the percentage of correct responses out of the total number of questions answered in that category, with scores ranging from 0 to 100. The change in pre/post scores was calculated by taking the differences in knowledge scores from baseline to pre-test, 10-days and 3 months survey.
Time Frame: baseline, pre-test (approximately 2-3 days after baseline), 10 days and 3 months
Population: Only participants who answered at least half of the knowledge questions for corresponding surveys were included in the analysis.
Measure: Mean (Standard Error); unit: Point
Groups:
- Arm II (Genomics Test Results, HOPE-Genomics): This group pools together Arm II and Arm III patients who have access to genomics test results from the HOPE-Genomics tool.
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) | Arm III (HOPE-Genomics, Genomics Test Results)
Number analyzed (Participants) | 139 | 140 | 139
Point
  Change from baseline to pre-test (approximately 2-3 days after baseline) | 2.76 (14.19) | 1.67 (13.36) | 7.39 (13.88)
  Change from baseline to 10 days: number analyzed (Participants) | 127 | 129 | 117
  Change from baseline to 10 days | 1.24 (16.92) | 4.86 (16.85) | 7.44 (16.95)
  Change from baseline to 3 months: number analyzed (Participants) | 115 | 121 | 111
  Change from baseline to 3 months | 1.63 (17.48) | 3.12 (18.59) | 6.04 (16.32)

ADVERSE EVENTS:
Time Frame: Since this is not a drug trial, there was no specific timepoint that was monitored for an adverse event to be recorded and patients were not assessed for specific adverse events. However, 19 patients died during the study, not due to study participation. The time frame where each participant was monitored/assessed for death was up till 9 months after their genetic testing.
Description: Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed. Please see above regarding adverse events.
Arm/Group | Arm I (Usual Care) | Arm II (Genomics Test Results, HOPE-Genomics) | Arm III (HOPE-Genomics, Genomics Test Results)
All-Cause Mortality (participants affected / at risk) | 6/155 | 8/155 | 5/155
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT04905082/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04905082/ICF_000.pdf